CLINICAL TRIAL: NCT03146702
Title: Evaluation of the Validity and Reliability of the Turkish Translation of The Emphasis-10 Questionnaire in Patients With Pulmonary Hypertension
Brief Title: Turkish Translation of The Emphasis-10 Questionnaire
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Pınar ÖDEVOĞLU, PT, MSc, Research Assistant, Istanbul University
Other Study IDs: TR-034
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Hypertension
Keywords: Quality of Life
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of Life — Patients self administor quality of life questionnaires such as Minnesota Living with Heart Failure Questionnaire and EmPHasis-10 questionnaire

SUMMARY:
Pulmonary Hypertension (PH) is a hemodynamic and physiopathological condition that is defined as an increase in mean pulmonary artery pressure ≥25 mmHg when measured at rest. PH often progresses to heart failure and premature deaths. PH is a progressive disease that has many causes, which can affect people of all ages, is characterized by shortness of breath, reduced exercise tolerance, psychological distress and tiredness and reduced quality of life. Surveys of SF-36, 'Nottingham Health Profiles' and 'Minnesota Life with Heart Failure' surveys are routinely performed in PH clinically. However, none of the questionnaires are specific to pulmonary hypertension, so they are incomplete in determining the condition of the disease and the patients. There is no Turkish questionnaire for patients with pulmonary hypertension and other surveys used are inadequate in determining the condition of the patient and the patient since they are not specific to the disease. The aim is to provide a Turkish questionnaire that is specific to pulmonary hypertension in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Pulmonary Hypertension
* Following at least 6 months of Pulmonary Hypertension policlinic
* Native Turkish
* People age 18 years or older

Exclusion Criteria:

* Those with cognitive impairment
* Those who have difficulty understanding or speaking Turkish

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Investigators include Pulmonary Hypertension patients who is following at least 6 months by the pulmonary hypertension policlinic. Patients had to be native turkish to newly translated EmPHasis-10 questionnaire to be valid. Patients who have cognitive impairment and difficulty understanding or speaking Turkish are excluded.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Validity | 8 months
  Validity of EmPHasis-10 Questionnaire
Reliability | 8 months
  Reliability of EmPHasis-10 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Odevoglu, MSc, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No